CLINICAL TRIAL: NCT05983705
Title: The Effect and Experience of the Brief Parental Program AFFEKT Within Primary Health Care - for Parents of Children With Externalizing Behaviors
Brief Title: The Effect and Experience of the Parental Program AFFEKT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Medtanken Group AB (Other); FoU i Västra Götalandsregionen (Unknown); Forte (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-01045; 2022-01045 (Other Grant/Funding Number: Swedish Resarch Council for Health, Working Life and Welfare); VGFOUREG-982199 (Other Grant/Funding Number: The Healthcare Committee, Region Västra Götaland)
Record Dates: First submitted 2023-07-03; First posted 2023-08-09 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Behavior, Child; Parenting; Parent-Child Relations; Stress; Quality of Life
Keywords: Randomized Controlled Trial; Qualitative Research; Parents; Child Behavior; Problem Behavior; Multicenter Study; Primary Health Care
MeSH Terms: conditions — Child Behavior; Problem Behavior | interventions — Aging

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial (RCT) and a qualitative study.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigators providing the psychoeducation and collecting the data at the information meeting (baseline) will be blinded since the randomization is carried out after that meeting and by an independent researcher.
  The individuals conducting the statistical analyses on the data from the RCT study will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment group (Experimental): The experiment group will receive written psychoeducation about children with externalizing behaviors, and start their parental program AFFEKT approximately one week from the information meeting (baseline).
  Interventions: Behavioral: AFFEKT - a manual based brief parent program for parents of children (aged 6-12 years) with externalizing behaviors.
- Control group (Active Comparator): The control group will receive written psychoeducation about children with externalizing behaviors, and start their parental program AFFEKT approximately seven weeks from the information meeting (when the experiment group has finished their AFFEKT program).
  Interventions: Behavioral: AFFEKT - a manual based brief parent program for parents of children (aged 6-12 years) with externalizing behaviors.

INTERVENTIONS:
Behavioral: AFFEKT - a manual based brief parent program for parents of children (aged 6-12 years) with externalizing behaviors. — The AFFEKT program includes five group sessions, two hours each, provided on a weekly basis. The program is delivered by therapist trained in Cognitive and Behavioral Therapy (CBT) and AFFEKT. The participants also receive a participation material, covering the same themes that are addressed in the program and working sheets for the home-assignments that are provided in-between sessions.

SUMMARY:
This project is the first to evaluate the effect and experience of the parent program AFFEKT, through a randomized controlled trial and qualitative study, within primary health care. The project will recruit 200 parents of children with externalizing behaviors, and evaluate the effect of AFFEKT and psychoeducation versus psychoeducation alone, on children's behaviors and mental health, and the parent's strategies and mental health. Through interviews the experience of AFFEKT will be investigated.

DETAILED DESCRIPTION:
Externalizing behaviors is a common problem among children. There are several parent programs for parents of children with externalizing behaviors, but many of these programs are time consuming. Within Medtanken Group AB a new brief parent program called AFFEKT has been developed. The clinical experience of the program has been promising, yet there are no previous randomized controlled trials or qualitative studies of AFFEKT.

The overall aim of this project is to examine the efficacy of the brief parenting program AFFEKT for parents of children with externalizing behaviors, and the parents experience of participating in AFFEKT. The project includes a quantitative study, including a randomized controlled trial (RCT), and a qualitative study.

Main aim and research question of the RCT part of the project:

The main aim of the RCT is to evaluate the efficacy of the brief parenting program AFFEKT. Is AFFEKT and psychoeducation targeting the parents more effective in changing the child's externalizing behaviors and mental health than psychoeducation alone? Primary research questions of the RCT

1. Will the outcome concerning the children's problematic behaviors improve statistically and significantly more in the experiment group (psychoeducation + AFFEKT) than in the control group (psychoeducation alone) post treatment?
2. Will there be statistical and significant effects of AFFEKT + psychoeducation on the children's problematic behaviors over time (6 and 12months after baseline)?

   Secondary research questions of the RCT
3. Will outcomes concerning the children's mental health improve statistically and significantly more in the intervention group (psychoeducation + AFFEKT) than in the control group (psychoeducation alone) post treatment?
4. Will the parental sense of competence, strategies, mental health, and quality of life have improved significantly more in the intervention group (psychoeducation + AFFEKT) than in the control group (psychoeducation alone)?
5. Will there be statistical and significant effects on the children's mental health, and the parent's sense of competence, strategies, mental health and quality of life over time (6 and 12months after baseline)?
6. Will changes in the parent's sense of competence, parental strategies, mental health and health-related quality of life mediate the changes in the child's externalizing behaviors and mental health over time?

Aim and specific research questions for the qualitative part of the study:

* The main aim of the qualitative study is to examine parents experience of the intervention AFFEKT, and how they perceive their child and relation to their child after the program.
* What aspects of AFFEKT did the parent's find helpful and what knowledge do the parents perceive that they have gained from their participation in AFFEKT? How do the parents perceive those previous situations they found difficult before the parental program AFFEKT, after participation? And what have changed in these situations?
* How has the parent's perception of the child changed, and in what way have the parent's relation to their child, changed after their participation in AFFEKT? Are there differences in the mothers and fathers' experiences of AFFEKT? The sample in both studies will be parents searching help for their children with externalizing behaviors, within the context of primary health care. The clinics that will be recruiting participants are all driven by Medtanken Group, but within different municipalities and counties in the Region of Västra Götaland, Sweden.

Sample size was determined after a power analysis, using G*Power. The power analysis used an effect size of 0.50, an alpha level of 0.05, and a power of 0.80. The number of patients needed was 64 in each group (experiment, control). With consideration to drop-outs N=200 will be recruited to the RCT. The qualitative study will include a random sample of 30 of these participants (15 women, 15 men).

Methods for data collection

All parents in contact with the clinics meeting the inclusion criteria will be asked to participate in the project. The parents willing to participate will be booked for a digital group information meeting through Microsoft Teams. These information meetings will be held after 10-14 families at one of the included clinics have shown interest in the project. At these meetings the parents will receive verbal and written information about the RCT and qualitative study and leave their written and informed consent. The participants will then answer the baseline questionnaires online, receive psychoeducation from a brochure and get a brief standardized information about AFFEKT.

After the information meeting (baseline) a psychologist within Medtanken Group (not part of the research group) will randomly assign the participants (single parents as one unit and couples as one unit) to either experiment or control group, using randomizerorg.se. The allocation ratio will be 1:1. Since the information meetings will be held consecutively at each clinic the randomization procedure will be consecutive as well.

The outcome measures are all answered by the parents. Data will be collected at baseline, pretreatment (+7 weeks) for the control group, post treatment (+6 weeks for the experiment group and +11 weeks for control group), +6 and +12 months. The questionnaires at baseline, +6 and +12 months will be online, and the questionnaires at the start and end of AFFEKT will be in paper and pen. The study participants will receive a gift certificate after they have finished their AFFEKT group and after they have completed the study.

The qualitative study will use semi-structured interview-guides. The participants who have agreed to be contacted for participation in an interview about their experiences of AFFEKT will be contacted 3 weeks after the last session and asked if they still would like to participate. Interviews will be conducted online, through Microsoft Teams or at the clinic where the participants received their treatment. The participants of the qualitative study will also receive a gift certificate.

Methods for data analyses

The RCT study will follow CONSORT standards. A participant flow-chart will be developed. For each group baseline demographics and characteristics will be presented. Data analyses will include both Intention to treat (ITT) and per protocol (PP) analyses, meaning the intended parents to treat and the once that completed the program and follow-up registrations will be analyzed separately. The level of statistical significance will be held at alpha 0.05. Bonferroni Corrections will be used to handle multiple analyses. The last-observation-carried-forward technique will be used for imputing missing values due to dropouts in the ITT analyses. Missing values on item level will be imputed with the mean value of that subscale for that respondent. Binary outcomes will be presented in both relative and absolute effect sizes. For each outcome estimated effect sizes and confidence intervals will be presented. Between group analyses will include baseline data, pre- and post-intervention data. Within group analyses will include baseline data, post-intervention data, 6month data and 12month data. Growth Curve Models will be performed to examine mean level stability and changes in parental outcomes using baseline data, post-intervention data, 6month data and 12month data. The twelve month follow up will not enable comparisons between groups, since all participants by then have received the intervention, however the sustainability of the results post intervention can be analyzed. Subgroup analyses will be based on parental gender, socio-economic status, and the age of the children. A drop-out analysis will also be conducted including both descriptive and analyzing statistics.

The material from the qualitative study and interviews will be transcribed and qualitative analyses such as thematic analysis and thematic reflexive analysis will be used to explore the research questions.

ELIGIBILITY:
Inclusion Criteria:

* Parent (or primary caregiver) to a child 6-12 years with externalizing issues
* Can communicate in Swedish

Exclusion Criteria:

* Attending other parental programs
* Non-communicable in Swedish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in disruptive behavior as assessed by the ECBI | The ECBI is measured at baseline for both groups, pre AFFEKT (+7 weeks) for the control group, post AFFEKT (+6 weeks) for the experiment group and (+11 weeks) for the control group, and at follow-up (+6 months and +1 year) for both groups.
  The Eyberg Child Behavior Inventory (ECBI; Eyberg & Ross, 1978) measures disruptive behavior problems in children through 36 items.

SECONDARY OUTCOMES:
Change in symptoms associated with ADHD as assessed by the SNAP-IV | The SNAP-IV is measured at baseline for both groups, pre AFFEKT (+7 weeks) for the control group, post AFFEKT (+6 weeks) for the experiment group and (+11 weeks) for the control group, and at follow-up (+6 and +1 year) for both groups.
  The Swanson, Nolan and Pelham Scale (SNAP-IV; Swanson et al., 1992) measures symptoms associated with ADHD in children. The Swedish version of the SNAP-IV includes 30 items (available at https://www.sfbup.se/wp-content/uploads/2020/04/SNAP-IV-SFBUP.pdf, the 27th of March, year 2022).
Symptoms and social deficits associated with autism spectrum disorders as assessed by the SRS-2 | The SRS-2 is measured at baseline for both groups.
  The Social Responsiveness Scale, second edition (SRS-2; Constantino & Gruber, 2012; Swedish version by Zander & Bölte) measures symptoms and social deficits associated with autism spectrum disorders through 65 items.
Change in global stress as assessed by the PSS -14 | The PSS is measured at baseline for both groups, pre AFFEKT (+7 weeks) for the control group, post AFFEKT (+6 weeks) for the experiment group and (+11 weeks) for the control group, and at follow-up (+6 months and +1 year) for both groups.
  The Perceived Stress Scale (PSS; Cohen, Kamarck & Mermelstein, 1983) measures global stress in adults. The Swedish version includes 14 items.
Change in general mental ill-health and health as assessed by the GHQ-12 | The GHQ-12 is measured at baseline for both groups, pre AFFEKT (+7 weeks) for the control group, post AFFEKT (+6 weeks) for the experiment group and (+11 weeks) for the control group, and at follow-up (+6 months and +1 year) for both groups
  The General Health Questionnaire (GHQ-12; Goldberg & Williams, 1988) measures self- rated general mental ill-health and health in adults through 12 items.
Change in quality of life as assessed by the BBQ | The BBQ is measured at baseline for both groups, pre AFFEKT (+7 weeks) for the control group, post AFFEKT (+6 weeks) for the experiment group and (+11 weeks) for the control group, and at follow-up (+6 months and +1 year) for both groups.
  The Brunnsviken Brief Quality of Life (BBQ; Lindner et al., 2016) measures subjective quality of life in adults through 12 items.
Treatment satisfaction as assessed by the CSQ-8 | The CSQ-8 is measured post AFFEKT (+6 weeks) for the experiment group and (+11 weeks) for the control group.
  The Client Satisfaction Questionnaire (CSQ-8; Nguyen, Attiksson and Stegner, 1983) is a questionnaire that measures treatment satisfaction through 8 items.

OTHER OUTCOMES:
Change in parental self-efficacy and parental satisfaction as assessed by the PSOC | The PSOC is measured at baseline for both groups, pre AFFEKT (+7 weeks) for the control group, post AFFEKT (+6 weeks) for the experiment group and (+11 weeks) for the control group, and at follow-up (+6 months and +1 year) for both groups.
  The Parenting Sense of Competence (PSOC; Johnston & Mash, 1989) measures parental self-efficacy (e.g., parents capability levels, problem-solving abilities and competence in their parental role) and parental satisfaction. The questionnaire consists of 16 items.
Change in the child's general health and health behaviors, and change in the parent's general health will be assessed by a questionnaire developed by the researchers | Measured at baseline, pre AFFEKT (+6 weeks) for the control group, post AFFEKT (+7 weeks ) for the experiment group and (+11 weeks) for the control group, and at follow-up (+6 months and +1 year) for both groups.
  In addition to the above established measurements, the questionnaire developed by the researchers measures the child's general health and health behaviors, and the parent's general health, through 10 single item questions.

CONTACTS AND LOCATIONS:
Overall Officials: Py Eriksson, Dr, Study Chair — Gothenburg University, Institute of Psychology
Locations (1):
- Medtanken Group AB, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Yes, there is a plan to make IPD supporting the results or analyses presented in published manuscripts available upon reasonable request. However, raw data (e.g., from the qualitative interviews) that contain personal information will not be shared, since it may lead to participant identification.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 3 months and ending 12 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. Proposals should be directed to the responsible researcher py.eriksson@psy.gu.se